CLINICAL TRIAL: NCT00937911
Title: YM150 Phase III Study - An Open-label, Multi-center Study in Subjects Undergoing Hip Fracture Surgery or Surgery in the Lower Extremities
Brief Title: Prevention of Venous Thromboembolism in Subjects Undergoing Hip Fracture Surgery or Surgery in the Lower Extremities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 150-CL-041
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Venous Thromboembolism
Keywords: YM150; Bleeding; Anticoagulant; Venous thromboembolism; FXa inhibitor
MeSH Terms: conditions — Venous Thromboembolism; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YM150 group (Experimental)
  Interventions: Drug: YM150

INTERVENTIONS:
Drug: YM150 — oral

SUMMARY:
The study objective is to evaluate the efficacy and safety of oral YM150 for prevention of venous thromboembolism in subjects undergoing hip fracture surgery or surgery in the lower extremities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing hip fracture surgery or patients undergoing surgery in the lower extremities other than hip fracture surgery
* Written informed consent obtained before screening

Exclusion Criteria:

* Subject has history of deep vein thrombosis and/or pulmonary embolism
* Subject has a hemorrhagic disorder and/or coagulation disorder
* Subject has had clinically important bleeding occurred within 90 days prior to the screening visit
* Subject has an acute bacterial endocarditis
* Subject has uncontrolled severe or moderate hypertension, retinopacy, myocardial infarction or stroke
* Subject is receiving anticoagulants/antiplatelet agents
* Subject has a body weight less than 40 kg

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Incidence of venous thromboembolism | Until day 12

SECONDARY OUTCOMES:
Incidence of deep vein thrombosis | Until day 35
Incidence of pulmonary embolism | Until day 35
All cause mortality | Until day 35
Incidence of bleeding event | Until day 35

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu
  - Shikoku
  - Tōhoku